CLINICAL TRIAL: NCT03718286
Title: Effects of Acute, Rapid Lowering of Low Density Lipoprotein Cholesterol With Alirocumab in Patients With ST Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Effects of Acute, Rapid Lowering of LDL Cholesterol With Alirocumab in Patients With STEMI Undergoing Primary PCI
Acronym: EPIC STEMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EPIC.STEMI.2018
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: ST Elevation Myocardial Infarction; Acute Coronary Syndrome; Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Physiological Effects of Drugs
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Acute Coronary Syndrome; Hypercholesterolemia; Hyperlipidemias; Dyslipidemias | interventions — alirocumab

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, sham-controlled parallel group clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alirocumab (Experimental)
  Interventions: Drug: Alirocumab
- Sham Control (Sham Comparator)
  Interventions: Other: Sham Control

INTERVENTIONS:
Drug: Alirocumab — 150 mg alirocumab administered prior to revascularization procedure, 2 weeks post-procedure and 4 weeks post-procedure.
  Arms: Alirocumab
Other: Sham Control — Sham injection prior to revascularization procedure, 2 weeks post-procedure and 4 weeks post-procedure.
  Arms: Sham Control

SUMMARY:
A randomized, double-blind, placebo controlled parallel group clinical trial evaluating the effects of acute treatment with a PCSK9 inhibitor (alirocumab) versus placebo on low-density lipoprotein (LDL) in 100 high-risk patients presenting with STEMI and referred for primary PCI.

The objective is to determine the effect of acute, rapid lowering of LDL cholesterol with alirocumab added to high dose statin therapy in patients with STEMI undergoing primary PCI. The hypothesis is that, in patients with STEMI undergoing primary PCI, rapid lowering of LDL cholesterol with a PCSK9 Inhibitor (alirocumab) initiated in the acute setting pre-PCI, will favourably affect LDL cholesterol concentrations compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with STEMI defined as both of the following: a) Symptoms of myocardial ischemia lasting for ≥ 30 minutes, and b) Definite ECG changes indicating STEMI: ST elevation of greater than 0.1 mV in two contiguous limb leads or 0.2 mV in two contiguous precordial leads.
* Referred for primary PCI for presenting symptoms.
* Randomized within 12 hours of symptom onset and prior to diagnostic angiography.

Exclusion Criteria:

* Age ≤18 years.
* Pregnancy or breastfeeding.
* Current or planned treatment with a PCSK9 inhibitor.
* Allergy or contra-indication to a PCSK9 inhibitor.
* Killip class ≥2.
* Known Creatinine clearance <30mL/min.
* Suspected takotsubo / stress-induced cardiomyopathy or acute pericarditis.
* Any other medical, geographic, or social factor making study participation impractical or precluding follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Percent change in direct LDL cholesterol | 6 weeks

SECONDARY OUTCOMES:
Percent change in Apo B | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shamir Mehta, MD MSc FRCPC, Principal Investigator — Population Health Research Institute; McMaster University
Locations (1):
- Hamilton Health Sciences, General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mehta SR, Pare G, Lonn EM, Jolly SS, Natarajan MK, Pinilla-Echeverri N, Schwalm JD, Sheth TN, Sibbald M, Tsang M, Valettas N, Velianou JL, Lee SF, Ferdous T, Nauman S, Nguyen H, McCready T, McQueen MJ. Effects of routine early treatment with PCSK9 inhibitors in patients undergoing primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: a randomised, double-blind, sham-controlled trial. EuroIntervention. 2022 Dec 2;18(11):e888-e896. doi: 10.4244/EIJ-D-22-00735. PMID 36349701